CLINICAL TRIAL: NCT03807960
Title: The Effect of Visual and Written Information Tools on Patient Controlled Analgesia Device Usage
Brief Title: Information for Patient Controlled Analgesia Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tuğba Karaman (Other)
Collaborators: Tokat Gaziosmanpasa University (Other)
Responsible Party: Sponsor-Investigator, Tuğba Karaman, Associate Professor,MD, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: pcı
Record Dates: First submitted 2019-01-11; First posted 2019-01-17 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Care; Hysterectomy; Health Communication
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- visual (Experimental): The video about patient controlled analgesia device (PCA) usage will shown to the patients via notebook.
  Interventions: Other: video
- written (Experimental): The written form which include the same knowledge will give to the patient for reading.
  Interventions: Other: written form
- control (Other): The anesthesiologist will describe the PCA usage as in the routine care to the control group patients.
  Interventions: Other: routine care

INTERVENTIONS:
Other: written form — The written form which include PCA usage information.
  Arms: written
Other: video — The video about PCA usage
  Arms: visual
Other: routine care — The routine description about PCA usage
  Arms: control

SUMMARY:
This study is aimed to show the effect of information method on properly usage of the patient controlled analgesia(PCA) device

DETAILED DESCRIPTION:
Postoperative pain is still a challenge for anesthesiologist. Patient controlled analgesia is an effective method for postoperative pain management. However, most of the patient can not use the device properly. The important cause of inabilities about device usage is insufficient information.In the patient information, visual, oral or written communication methods can be chosen. However, which method is suitable for our patient group is not clear.This study is aimed to show the effect of information method on properly usage of the patient controlled analgesia(PCA) device

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* Elective hysterectomy

Exclusion Criteria:

* Opioid abuse or Chronic opioid usage
* opioid allergy
* obesity(BMI>30)
* psychiatric disease
* more than American Anesthesiologist Score 2

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Pain Score | At postoperative 24th hours.
  Numeric rating scale (0 to 10) will be used for postoperative pain score

SECONDARY OUTCOMES:
Postoperative analgesic consumption | Up to the postoperative 24th hours.
  Total opioid dosage will be recorded
PCA device usage | During postoperative 24 hours
  The number of demand dose
PCA device demand dose duration | During postoperative 24hours
  The duration of the patients' demanding dose
Patient's satisfaction | At the postoperative 24th hours
  The numeric rating scale (0 to 10) will be used. In this scale 0 will be the worst, 10 will be the best satisfaction.
The change of the postoperative pain score | Up to the postoperative 24th hours.
  Numeric rating scale (0 to 10) will be used to evaluate the pain score. The change in this score during postoperative 24 hours will be calculated.(the first score will be extracted from the last score)

OTHER OUTCOMES:
Length of stay hospital | Up to the postoperative 10 days
  Number of the day that patients stay at hospital will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Karaman, MD, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University Hospital, Tokat Province, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided